CLINICAL TRIAL: NCT02148393
Title: Elective Blastocyst Vitrification for Endometrial Receptivity Enhancement in High-responder Patients Undergoing in Vitro Fertilisation/Intracytoplasmatic Sperm Injection (IVF/ICSI)
Brief Title: Implantation Enhancement by Elective Cryopreservation of All Viable Embryos
Acronym: ICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Samuel Santos-Ribeiro, M.D., Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-128; 2014-001480-12 (EudraCT Number)
Record Dates: First submitted 2014-05-16; First posted 2014-05-28 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Infertility; OHSS
MeSH Terms: conditions — Infertility | interventions — Vitrification; Parturition; Chorionic Gonadotropin; Utrogestan; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): In the control group, following oocyte retrieval, intensified luteal phase support for fresh embryo transfer (with Pregnyl®, Utrogestan® and Progynova®) will be performed. Fresh ET in the uterine cavity will be performed on the 5th day of embryo development at blastocyst stage under ultrasound guidance whenever possible.
  Interventions: Procedure: Intensified luteal phase support for fresh embryo transfer; Drug: Pregnyl®; Drug: Utrogestan®; Drug: Progynova®
- Intervention (Experimental): Elective vitrification with subsequent-cycle embryo thawing/transfer (CryoBioSystem®) will be performed. Hence, no luteal phase support will be provided immediately after oocyte retrieval. Instead, patients will wait for a subsequent cycle before starting exogenous hormone therapy for endometrial preparation.
  On the day of embryo transfer, blastocyst(s) will be warmed one by one until one or two blastocysts are suitable for transfer. ET to the uterine cavity will be performed under ultrasound guidance whenever possible.
  Interventions: Procedure: Vitrification with subsequent-cycle embryo thawing/transfer; Device: CryoBioSystem®

INTERVENTIONS:
Procedure: Vitrification with subsequent-cycle embryo thawing/transfer — The vitrification process will be performed under the same conditions of all other vitrification procedures usually performed in our centre. In summary, vitrification will be accomplished using closed high security straws (CryoBioSystem®) in combination with dimethylsulfoxide, ethylene glycol and sucrose as cryoprotectants (Irvine ScientificR Freeze Kit®).
  In the meantime, patients will wait for a subsequent cycle before starting exogenous hormone therapy for endometrial preparation.
  Arms: Intervention
Procedure: Intensified luteal phase support for fresh embryo transfer — A single administration of 1500 IU of exogenous hCG (Pregnyl®) 1 hour after oocyte retrieval followed by daily vaginally-administered progesterone 200 mg tid (Utrogestan®) and oestradiol valerate 2 mg bid (Progynova®).
  Arms: Control
Drug: Pregnyl® — 1500 IU
  Other Names: hCG
  Arms: Control
Drug: Utrogestan® — 200 mg tid
  Other Names: Vaginal progesterone
  Arms: Control
Drug: Progynova® — 2 mg bid
  Other Names: Estradiol valerate
  Arms: Control
Device: CryoBioSystem® — CryoBioSystem® in combination with dimethylsulfoxide, ethylene glycol and sucrose as cryoprotectants (Irvine ScientificR Freeze Kit®) closed in high security straws
  Arms: Intervention

SUMMARY:
A randomised controlled open-label clinical trial to compare the clinical pregnancy rates between fresh embryo transfer and elective all-embryo vitrification with thawing and transfer in a subsequent cycle in high-responders

DETAILED DESCRIPTION:
Two-arm randomised, single-centre, controlled open-label trial. Summarily, women undergoing exogenous gonadotropin ovarian stimulation for ART in a gonadotropin-releasing hormone (GnRH) antagonist down-regulated cycle and at high risk for ovarian hyperstimulation syndrome (OHSS) will be included in either the control ("fresh embryo transfer") or intervention ("subsequent vitrified-warmed embryo transfer") groups. Women in the control group will undergo GnRH agonist triggering followed by intensified luteal phase support while the intervention group will electively vitrify all viable embryos after GnRH triggering and perform the embryo transfer (ET) in a subsequent unstimulated cycle.

Ovarian stimulation, ultrasound and hormonal monitoring, ovulation induction, oocyte retrieval, embryology procedure, IVF and luteal support will be according to how they are normally performed in our centre.

All women included will undergo artificial ovarian stimulation with GnRH antagonist down-regulation with daily injections of either ganirelix (Orgalutran®) or cetrorelix (Cetrotide®). Treating physicians will opt on which exogenous gonadotropins should be used according to the patient's profile and preference and can include either recombinant follicle stimulating hormone (FSH) or highly purified urinary human menopausal gonadotropin (HP-HMG). Ovarian stimulation will commence after it is confirmed that the patient is not pregnant and has basal levels of oestradiol, progesterone, FSH and luteinising hormone (LH). The stimulation will be monitored simultaneously by pelvic ultrasound and hormonal analyses (oestradiol, progesterone), starting on day 7 of stimulation and then every 1 to 3 days, according to the individual endocrine profile and follicular development.

Final oocyte maturation will be triggered with 0.2 mg triptorelin (Decapeptyl®, Gonapeptyl®) as soon as 3 follicles of ≥17 mm are observed. A GnRH agonist will be the preferred triggering agent for both groups to reduce the risk of severe OHSS associated with human chorionic gonadotropin (hCG) triggering in high-responders. Oocyte retrieval will be performed 36 hours after hCG administration under either local anaesthesia with analgesic premedication or general anaesthesia, according to patient preference.

IVF/ICSI will be performed, using the specimen of sperm made available by the male progenitor on the day of oocyte retrieval.

The choice to transfer one or two embryos will be decided by the clinician at consultation mainly depending on the patient's age and the number of embryos replaced in the previous treatment cycles, according to Belgian law.

ELIGIBILITY:
Inclusion Criteria:

* First or second IVF/ICSI cycle
* High response to ovarian stimulation (defined as presence of ≥18 follicles of ≥11 mm on the day of GnRH triggering)
* GnRH antagonist down-regulation
* Signed informed consent
* Patients can be included only once in the trial
* Planned replacement of 1 or 2 blastocysts

Exclusion Criteria:

* Other known reasons for impaired implantation (i.e. hydrosalpinx, fibroid distorting the endometrial cavity, Asherman's syndrome, thrombophilia or endometrial tuberculosis)
* Oocyte/embryos donation acceptors
* Embryos planned to undergo preimplantation genetic diagnosis/screening
* Body mass index ≥35 or ≤18
* Women who have previously enrolled in the trial
* Those unable to comprehend the investigational nature of the proposed study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 212 (Actual)
Dates: Start 2014-05; Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rates | 7 weeks
  Pregnancy visible under transvaginal pelvic ultrasound

SECONDARY OUTCOMES:
Ovarian hyperstimulation syndrome incidence | 8 weeks
  Observation of early-onset ovarian hyperstimulation syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Santos-Ribeiro, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Christophe Blockeel, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Lisboa, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zaat T, Zagers M, Mol F, Goddijn M, van Wely M, Mastenbroek S. Fresh versus frozen embryo transfers in assisted reproduction. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD011184. doi: 10.1002/14651858.CD011184.pub3. PMID 33539543
- [Derived] Santos-Ribeiro S, Mackens S, Popovic-Todorovic B, Racca A, Polyzos NP, Van Landuyt L, Drakopoulos P, de Vos M, Tournaye H, Blockeel C. The freeze-all strategy versus agonist triggering with low-dose hCG for luteal phase support in IVF/ICSI for high responders: a randomized controlled trial. Hum Reprod. 2020 Dec 1;35(12):2808-2818. doi: 10.1093/humrep/deaa226. PMID 32964939